CLINICAL TRIAL: NCT05753891
Title: Trapeziectomy With Internal Brace Versus Ligament Reconstruction With Tendon Interposition; a Prospective Study
Brief Title: Trapeziectomy: Internal Brace vs. Ligament Reconstruction (Prospective)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Charles S Day, Interim Chairman & Medical Director, Professor of Orthopaedic Surgery, Department of Orthopaedic Surgery & Service Line, Wayne State University School of Medicine, Henry Ford Health, Henry Ford Health System
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16162
Record Dates: First submitted 2023-02-23; First posted 2023-03-03 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Basilar Thumb Arthritis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Carpometacarpal (CMC) Suture Tape Ligament Reconstruction (Experimental): Patients in this arm will undergo trapeziectomy with suture tape suspension of the 1st metacarpal to the 2nd metacarpal via Arthrex InternalBrace device. This is the experimental group.
  Interventions: Device: Suture Tape Reconstruction
- Carpometacarpal (CMC) Standard Ligament Reconstruction (No Intervention): Patients in this arm are considered the control group and will undergo trapeziectomy with ligament reconstruction and tendon interposition.

INTERVENTIONS:
Device: Suture Tape Reconstruction — This intervention will utilize a suture tape to suspend the 1st and 2nd metacarpal post trapeziectomy compared to the standard procedure of a trapeziectomy followed by ligament reconstruction and tendon interposition.
  Other Names: Arthrex InternalBrace
  Arms: Carpometacarpal (CMC) Suture Tape Ligament Reconstruction

SUMMARY:
This study seeks to compare two methods of trapeziectomy for basilar thumb arthritis. The first is trapeziectomy with ligament reconstruction and tendon interposition, which means removing the trapezium bone and filling the void with a tendon graft. This is the most commonly used procedure and the control group. The experimental group is trapeziectomy with suture tape suspension of the 1st metacarpal to the 2nd metacarpal. This is using a device called the InternalBrace, produced by Arthrex.

ELIGIBILITY:
Inclusion Criteria:

* Patients of Henry Ford Orthopedic Service Line
* Symptomatic basilar thumb arthritis refractory to conservative management

Exclusion Criteria:

* Significant medical comorbidity precluding safe surgery, as determined by the operating surgeon. This may include cardiac disease, renal disease, liver disease, pulmonary disease, or heavy substance abuse.
* Requirement for additional procedures at the 1st carpometacarpal joint, including trapezoid excision-whole or partial-or metacarpal osteotomy. Of note other existing conditions requiring intervention on a separate surgical site such as concomitant carpal tunnel syndrome or trigger fingers will NOT be used as exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Pinch Strength | 6 months post procedure
  Pinch Strength measurements

SECONDARY OUTCOMES:
PROMIS-UE | 6 months post procedure
  Patient-Reported outcomes measurement information system (PROMIS) Upper Extremity (UE) item bank to record upper extremity function.

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States